CLINICAL TRIAL: NCT01315054
Title: A Methadone Maintenance Treatment Outcome Study in Three Provinces in China: Comparative Evaluation of the Impact of an Intensive Health Care Provider Training Program
Brief Title: A Methadone Maintenance Treatment Outcome Study in Three Provinces in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDC-CGH-6014; CN_09_217 (Other Grant/Funding Number: OGAC)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: HIV; Hepatitis C; Syphilis; Herpes Simplex Type II
Keywords: IDUs; high risk behaviors; HIV; MMT dosage and retention; psychosocial services
MeSH Terms: conditions — Hepatitis C; Syphilis | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control arm (Other): Using currently practiced methadone dosage prescription methods
  Interventions: Other: national guidelines
- MMT provider dosage training (Experimental): Intensive health care provider training on prescribing methadone dosage based on national guidelines
  Interventions: Behavioral: MMT provider dosage training; Other: national guidelines
- MMT provider dosage training/counseling (Experimental): Intensive health care provider training on prescribing methadone dosage, plus providing on-site psychosocial counseling services and peer support to clients .
  Interventions: Behavioral: MMT provider dosage training; Behavioral: targeted counseling; Other: national guidelines

INTERVENTIONS:
Behavioral: MMT provider dosage training — Training on methadone dosing provided to health care providers working in methadone maintenance clinics
  Other Names: training
  Arms: MMT provider dosage training; MMT provider dosage training/counseling
Behavioral: targeted counseling — targeted counseling provided to methadone maintenance clinic attendees
  Other Names: counseling
  Arms: MMT provider dosage training/counseling
Other: national guidelines — Provided a hard copy of the existing national guidelines for methadone dosing
  Other Names: dosing guidelines

SUMMARY:
The primary goal of this PHE is to determine the effectiveness of a tailored education program for MMT service providers. It was to be evaluated through methadone dose levels prescribed to new patients after training completion. The effects of methadone dose, with and without the inclusion of additional counseling services, would be measured through MMT retention and illicit opioid use.

DETAILED DESCRIPTION:
Methadone treatment has became one of main actions taken in China to control the spread of HIV among drug users. However，the average methadone dose used is relatively low. An intensive methadone maintenance treatment (MMT) provider training on methadone dosage may be effective in increasing the methadone dose levels prescribed to new patients. The study will evaluate the effectiveness of a tailored education program for MMT service providers using subsequent methadone dose prescribed to new patients. The effects of methadone dose, with and without the inclusion of additional psychosocial services, will then be measured through MMT retention and illicit opioid use.

ELIGIBILITY:
Inclusion Criteria:

* client participants will include both men and women who are opiate-dependent drug users who started MMT not more than one month prior to enrollment in the study
* 18 years of age or older
* residing in the study areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4258 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
MMT retention rate | 12 months
  % of patients retained at the end of the year after Methadone maintenance treatment
Illicit opioid use rate | 12 months
  by urinalysis and self-report

SECONDARY OUTCOMES:
HIV, HCV, syphilis and HSV-2 infection seroconversion rate | 12 months
  Patients who were negative converted to being seropositive
High risk needle practice | 12 months
  Shared needles used for drug injections without cleaning procedures involved
High risk sexual practice | 12 months
  Sex without condoms and also with multiple partners
Quality of life（WHO Quality of Life -BREF） | 12 months
  Scale of quality of life by WHO
All-cause mortality | 12 months
  Patients die by all causes during the program

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bulterys, MD, PhD, Principal Investigator — US CDC GAP China
Locations (1):
- National Center for HIV/STD Prevention and Control, China CDC, Beijing, China